CLINICAL TRIAL: NCT06839430
Title: Therapeutic Effect of Using Injectable Hypertonic Saline 5% Versus Injectable Dextrose 20% on Pain in Painful Cases of Disc Displacement with Reduction ( a Randomized Clinical Trial)
Brief Title: Therapeutic Effect of Using Injectable Hypertonic Saline 5% Versus Injectable Dextrose 20% on Pain in Painful Cases of Disc Displacement with Reduction
Acronym: RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Allah Gamal Salah, Aya Allah Gamal, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: injection in TMJ
Record Dates: First submitted 2025-02-17; First posted 2025-02-21 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: TMJ Disc Displacement with Reduction
MeSH Terms: interventions — Saline Solution, Hypertonic; Sodium Chloride

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- painful cases with disc displacement with reduction (Active Comparator)
- painful cases of disc displacement with reduction (Experimental)
  Interventions: Other: hypertonic saline 5% sodium chloride

INTERVENTIONS:
Other: hypertonic saline 5% sodium chloride — Hypertonic saline acts as an analgesic by alleviating nociceptive pain from inflamed tissues, which may include bone, connective tissue , synovium , or a combination of these Hypertonic saline results in safe and remarkable outcomes on knee pain, stiffness and function compared with intra-articular dextrose injection
  Arms: painful cases of disc displacement with reduction
Other: hypertonic dextrose 20% — A recent study showed the sensorineural analgesic effect of 5% dextrose prolotherapy in the treatment of chronic low back pain ,Therefore, the mechanism of action for dextrose prolotherapy is hypothesized to work through reducing peripheral sensitization and targeting structural dysfunction

SUMMARY:
This study is aiming to assess effect of hypertonic saline 5% in comparison to dextrose 20% on pain ,inter-insical opening and movements of jaw in painful cases of disc displacement with reduction

DETAILED DESCRIPTION:
Intra-articular disorders of the TMJ have been defined as an abnormal positional relationship between the disc and the condyle, articular eminence, and/or articular fossa.

The term internal derangement of the temporomandibular joint (TMJ) indicates an abnormal relationship between the disc, the condyle, and the articular eminence that constrains proper joint function

The disc displacement could be with or without reduction. In disc displacement with reduction, the disc is displaced anterior to the condylar head and remains in this position as long as the mouth is closed. Upon mouth opening, the disc regains its position on the condylar head. The movement of the disc onto and off the condylar head may lead to a clicking sound .

The precise source of internal derangements is not clear; however, it is a complex disorder likely caused by a combination of micro- or macro-trauma, parafunctional behavior, laxity of the joint's soft tissues, and alterations in the synovial fluid's composition

The aims of the internal derangement treatment include alleviating pain, reducing or eliminating joint noises, increasing the degree of mouth opening, and consequently restoring normal TMJ function.

Soft diet, behavior adjustment, analgesics, occlusal splints, intra-articular injections, physiotherapy, arthrocentesis, arthroscopy, and open joint surgery are the most common therapeutic techniques Injecting a non pharmacological irritant solution ,such as dextrose, into the area of the tendons or ligaments is known as prolotherapy, which is also known as regenerative injection therapy. It is hypothesized that this procedure elicits a non inflammatory or inflammatory process that ultimately leads to the deposition of new collagen fibers that strengthen lax tendons or ligaments and possibly encourage the release of local growth factor Different substances have been utilized for prolotherapy, but hypertonic dextrose is the most commonly utilized solution since it is affordable, accessible, and safe to inject Dextrose solution has been used at various concentrations ranging from 10% to 50% The superior joint space and peri-capsular soft tissues are usually injected during traditional prolotherapy of the TMJ.

Injection treatment of TMJs is currently one of the recognized therapeutic techniques.

Due to its invasive nature, only patients who have exhausted the less invasive treatment options are typically eligible for injection treatment.

Depending on the injectable substance used, injection treatment provides pain relief and increases the range of mandibular mobility Hypertonic saline , administered via intra-articular injection has been widely used in many previous clinical trials ,it has been used in patients with knee osteoarthritis and show significant improvement regarding pain, stiffness and function of joint hypertonic saline has a significant pain relief effect ,it acts as an analgesic by alleviating nociceptive pain from inflamed tissues, which may include bone, connective tissue, synovium, or a combination of these

ELIGIBILITY:
Inclusion Criteria:

* presence of one or more of the following observations in one or both temporomandibular joints:

  1. pain.
  2. audible clicking.
  3. mandibular deviation on opening.
  4. Failure of conservative treatment

Exclusion Criteria:

* The clinical or radiographic signs of disc displacement without reduction, osteoarthritis, or articular bony changes.

  * Previous TMJ surgery, arthrocentesis, , or the presence of any systemic disease that would affect the TMJ anatomy or mechanical function.
  * A history of allergic reactions to any components of the injectable solution.
  * Infection of the affected joint and pre-auricular area.
  * Previous surgery of the affected joint

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2026-08-20 (Estimated); Study Completion 2026-09-20 (Estimated)

PRIMARY OUTCOMES:
Severity of pain | baseline and at 6 months
  severity of pain is measured by Visual analog scale (VAS) From (0-10) Where 0: no pain 10: worst pain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gibaly A, Abdelmoiz M, Alghandour AN. Evaluation of the effect of dextrose prolotherapy versus deep dry needling therapy for the treatment of temporomandibular joint anterior disc displacement with reduction: (a randomized controlled trial). Clin Oral Investig. 2024 Aug 8;28(9):475. doi: 10.1007/s00784-024-05830-z. PMID 39115583
- [Background] Mohammed MR, Hamad SA, Al-Dawoody AD, Shehab AA, Ahmed OS. Effect of dextrose prolotherapy on internal derangement of the temporomandibular joint. Eur Rev Med Pharmacol Sci. 2023 Jun;27(11):4883-4889. doi: 10.26355/eurrev_202306_32605. PMID 37318462
- [Background] Zin'kovskii VG, Golovenko NIa, Bogatskii AV. [Nature of the relation between the anticonvulsant action of phenazepam and its concentration in mouse brain]. Biull Eksp Biol Med. 1981;91(1):40-2. Russian. PMID 7214004